CLINICAL TRIAL: NCT01509248
Title: Population Pharmacokinetics and Metabolomic Analysis of Aminopylline/Theophylline Drug Levels in Preterm Infants With Apnea of Prematurity
Brief Title: Population Pharmacokinetics and Metabolomics of Theophylline in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Seoul National University Boramae Hospital (Other); Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Han-Suk Kim, Associate Professor & Director of Neonatal Intensive Care Unit, Seoul National University Hospital
Other Study IDs: TP-PopPK-Metabol
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Apea of Prematurity
Keywords: Theophylline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
1. Population pharmacokinetics : The purpose of this study is

   - to investigate the population pharmacokinetics of theophylline in premature Korean infants and to assess the influence of demographic and clinical covariates.
2. Metabolomics : The purpose of this study are

   * to predict serum theophylline levels and to assess CYP1A2 activities in premature infants by analyzing urinary metabolites of theophylline
   * to examine which factors affect clearance of theophylline and CYP1A2 activity in premature infants

ELIGIBILITY:
Inclusion Criteria:

* Inborn preterm infants (GA < 37 weeks)
* Dx : Apnea of prematurity
* Tx : Aminophylline / Theophylline
* Informed consent of parents

Exclusion Criteria:

* Major congenital anomaly
* Expired within 72 hours
* Proven secondary apnea

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Admitted to Neonatal Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2010-05

REFERENCES:
- [Derived] Kim SE, Kim BH, Lee S, Sohn JA, Kim HS, Cho JY, Yoon SH, Jang IJ, Yu KS, Lim KS. Population pharmacokinetics of theophylline in premature Korean infants. Ther Drug Monit. 2013 Jun;35(3):338-44. doi: 10.1097/FTD.0b013e3182866695. PMID 23666573